CLINICAL TRIAL: NCT05124691
Title: An Adaptive Phase II/III SingleBlinded, Randomized, MultiCentre, ParallelGroup, Active Controlled, Superiority Study to Evaluate the Safety and Efficacy of a Single Day or 3day Single Dose of an ALBENDAZOLE IVERMECTIN Coformulation vs ALBENDAZOLE for the Treatment of SoilTransmitted Helminth Infections (Trichuris Trichiura, Hookworm, Strongyloides Stercoralis) in Paediatric and Young Adult Population
Brief Title: Evaluation of Effectiveness of ALBENDAZOLIVERMECTIN Coformulation vs ALBENDAZOLE for Treatment of Intestinal Worms
Acronym: ALIVE
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Primary Endpoint met
Sponsor: Barcelona Institute for Global Health (Other)
Collaborators: Leiden University Medical Center (Other); Bahir Dar University (Other); Centro de Investigacao em Saude de Manhica (Other); London School of Hygiene and Tropical Medicine (Other); Kenya Medical Research Institute (Other); Laboratorios Liconsa (Industry); Universidad de León (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALIVE
Record Dates: First submitted 2021-11-16; First posted 2021-11-18 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Helminthes; Infestation, Intestinal
Keywords: soil-transmitted helminths; pediatric; adult; albendazole; ivermectin; coformulation
MeSH Terms: conditions — Helminthiasis | interventions — Albendazole; Ivermectin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Albendazole (Active Comparator): Albendazole 400 mg single dose
  Interventions: Drug: Albendazole
- FDCx1. Albendazole and Ivermectin Fixed Dose Coformulation (Experimental): Single dose of a tablet of FDC 400mg18mg or 400mg9mg. (i) For participants <45 kg of body weight at baseline: FDC of 400mg ALB 9mg IVM. (ii) For participants ≥45 kg of body weight at baseline: FDC of 400mg ALB18mg IVM
  Interventions: Combination Product: Albendazole and Ivermectin fixed dose coformulation
- FDCx3. Albendazole and Ivermectin Fixed Dose Coformulation 3 days (Experimental): Daily dose of a tablet of FDC 400mg18mg or 400mg 9mg for 3 days. (i)For participants <45 kg of body weight at baseline: FDC of 400mg ALB9mg IVM. (ii) For participants ≥45 kg of body weight at baseline: FDC of 400mg ALB 18mg IVM.
  Interventions: Combination Product: Albendazole and Ivermectin fixed dose coformulation

INTERVENTIONS:
Combination Product: Albendazole and Ivermectin fixed dose coformulation — 400 mg Albendazole - 9 mg Ivermectin OR 400 mg Albendazole - 18 mg Ivermectin
  Arms: FDCx1. Albendazole and Ivermectin Fixed Dose Coformulation; FDCx3. Albendazole and Ivermectin Fixed Dose Coformulation 3 days
Drug: Albendazole — Albendazole 400mg single dose
  Arms: Albendazole

SUMMARY:
The purpose of this clinical trial is to evaluate a fixed-dose co-formulation (FDC) of ivermectin and albendazole for the treatment of all Soil Transmitted helminths (STH). The current strategy to control STH in endemic areas is mass administration of albendazole or mebendazole, mainly to pre-school and school-aged children.

Although this treatment works well for some STH species, efficacy against Trichuris trichiura is poor and it is not effective Strongyloides stercoralis. Thus new drugs or drug combinations are an urgent priority to increase the effectiveness of control programmes. Furthermore, the World Health Organisation has recommended combination therapy of ivermectin with albendazole. The trial proposed, is an adaptive phase II/III trial where the phase II component will evaluate the safety of the FDC as a single dose or 3-day single dose regimen for the treatment of T. trichiura in paediatric population. After analysis of the safety results the phase III trial will be executed to evaluate the efficacy of the FDC as a single dose or 3-day single dose regimen compared to the standard single dose regimen of ALB (400 mg) for the treatment of T. trichiura, hookworm and S. stercoralis in paediatric and young adult population. The estimated total sample size for the adaptive design (phase II and III component) is 1223 participants. Of these, 126 will be enrolled in the phase II and 1097 in the phase III components respectively in an adaptive trial design.

DETAILED DESCRIPTION:
An adaptive phase II/III clinical trial to evaluate the Safety and Efficacy of a Single Day or 3-day Single Dose of an ALBENDAZOLE-IVERMECTIN Coformulation vs ALBENDAZOLE for the Treatment of Soil-Transmitted Helminth Infections. The estimated total sample size for the adaptive design (phase II and III components) is 1223 participants. Of these, 126 will be enrolled in the phase II and 1097 in the phase III components.

Phase II component (Kenya only)

Unicentric, 3-arm, parallel, open-label, individually randomised, phase II trial to determine in three weight groups, the safety of the ALBENDAZOLEIVERMECTIN Co-formulation given as a Single Day or 3-day Single Dose regimen for the treatment of Trichuris trichiura in children and young adult aged between 5 to 18 years. Estimated sample size: 126 participants Participants will be stratified in three different weight groups in order to gradually increase the dose of ivermectin in the Fixed Dose Co-formulation (FDC):

* Group 1 (38 participants): with body weight of 23-<30 Kg will receive 300-391 µg/Kg IVM (FDC 400mg-9mg) or ALB
* Group 2 (38 participants): with body weight of 30-45 Kg will receive 400-600 µg/Kg IVM (FDC 400mg-18mg) or ALB.
* Group 3 (50 participants): with body weight of 15-23 Kg will receive 391-600 µg/Kg IVM (FDC 400mg-9mg) or ALB. Where FDC stands for Fixed Dose Co-formulation and ALB stands for Albendazole. Then, the participants will be allocated to one of the three study arms with unequal probability (ALB: p=0.2, n=26; FDCx1: p=0.4, n=50; FDCx3: p=0.4, n=50) starting with group 1.

  * Treatment Arm 1: Single dose of a tablet of ALBENDAZOLE 400 mg (active control arm).
  * Treatment Arm 2: Single dose of a tablet of ALBENDAZOLEIVERMECTIN Co-formulation.
  * Treatment Arm 3: Daily dose of a tablet of ALBENDAZOLE-IVERMECTIN Co-formulation for 3 consecutive days.

Phase III Component

A multi-centre, 3-arm, parallel, open-label, randomised, phase III trial to compare safety and efficacy of the active control arm (current standard of care) against 2 experimental arms for the treatment of T. trichiura, hookworm and S. stercoralis, in children and young adult aged between 5-18 years in three subSaharan African countries (Ethiopia, Kenya and Mozambique) We hypothesise that the FDC of Ivermectin (IVM) and ALB either at single or 3- day regimens will be more effective against some species of Soil Transmitted Helminths (STH) (T. trichiura, hookworm and S. stercoralis) compared to the current use of a single dose regimen of 400mg ALB. Estimated sample size: 1097 participants Participants will be randomly allocated with unequal probability, according to the specific expected cure rate by treatment and specie, to one of the three study treatment arms.

* Treatment Arm 1: Single dose of a tablet of ALB 400 mg (active control arm).
* Treatment Arm 2: Single dose of a tablet of FDC 400mg-18mg or 400mg-9mg.

  * For participants <45 kg of body weight at baseline: FDC of 400mg ALB- 9mg IVM.
  * For participants ≥45 kg of body weight at baseline: FDC of 400mg ALB-18mg IVM.
* Treatment Arm 3: Daily dose of a tablet of FDC 400mg-18mg or 400mg9mg for 3 days.

  * For participants <45 kg of body weight at baseline: FDC of 400mg ALB-9mg IVM.
  * For participants ≥45 kg of body weight at baseline: FDC of 400mg ALB- 18mg IVM.

In the phase III component, allocation of participants to study arms will be done by block randomization and stratified by the species of STH. Treatment allocation for each study participant will be concealed in opaque sealed envelope that will be opened only after enrolment. Study participants will be assigned a unique number linked to the allocated treatment group.

The phase II and III trial components comprise of a screening phase, an enrolment phase, a treatment phase, a post-treatment phase with follow-up visits, and early withdrawal/end-of-study evaluations. Participants recruited in Mozambique will be offered to be tested for HIV serostatus due to the high HIV prevalence in the country, but the result will not determine the participant's eligibility. In Kenya and Ethiopia, the low HIV prevalence does not justify HIV testing

ELIGIBILITY:
Inclusion Criteria:

* Positive infection test by microscopy for at least one of the following STH: T. trichiura, hookworms and/or larvae of S. stercoralis.
* Weight ≥15 Kg.
* Male or female, aged 5 to 18 years.
* Female participants who are ≥12 years old (or female post menarche) must have a negative urine pregnancy test at screening or at the time of randomization.
* Ability to take oral medication and willingness to comply with all study procedures.
* Parental acceptance to participate in the study by obtaining a signed and dated informed consent form approved by the Regulatory authorities. In addition, verbal assent will be obtained from children aged 12-18 years.

Exclusion Criteria:

* Intake of ALB, mebendazole and/or IVM, or any potentially interacting drug three months before screening.
* Residence outside the study area or planning to move away in the four weeks following recruitment.
* Epidemiological risk of infection by Loa loa.
* Serious medical illness, per investigator's criteria.
* Any participant's condition that would prevent the appropriate evaluation and followup, as per investigator's criteria.
* Known hypersensitivity to any components of either of the study treatment.
* Positive pregnancy urine test, pregnant or first week postpartum.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1001 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Munoz, MD, PhD, Principal Investigator — Barcelona institue for Global health
Locations (3):
- Bahir Dar University, Colleges of Medicine and Health Sciences (BDU-CMHS), Bahir Dar, Ethiopia
- Kenya Medical Research Institute (KEMRI), Nairobi, Kenya
- Centro de Investigação em Saúde da Manhiça (CISM), Manhiça, Maputo Province, Mozambique

IPD SHARING:
Plan to Share IPD: Yes
All data from the ALIVE clinical trial (phase II and phase III) have been upload to the Infectious Diseases Data Observatory (IDDO). IDDO is a scientifically independent, multi-disciplinary coalition of the global infectious disease and emerging infections communities. Thus, data will be available upon request in a collaborative data repository for verification and re-use.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data is already available upon request to IDDO
Access Criteria: All data sharing request received by IDDO will be addressed to the project consortium members who will approve/reject the data sharing based on the relevance of the proposal.
URL: https://www.iddo.org/

REFERENCES:
- [Derived] Krolewiecki A, Kepha S, Fleitas PE, van Lieshout L, Gelaye W, Messa A Jr, Gandasegui J, Algorta J, Novela V, de Jesus A, Rono M, Degarege D, Bedane D, Mwahanje J, Mandomando I, Mwandawiro C, Enbiale W, Munoz J; Stopping Transmission of Intestinal Parasites (STOP) consortium. Albendazole-ivermectin co-formulation for the treatment of Trichuris trichiura and other soil-transmitted helminths: a randomised phase 2/3 trial. Lancet Infect Dis. 2025 May;25(5):548-559. doi: 10.1016/S1473-3099(24)00669-8. Epub 2025 Jan 10. PMID 39805305
- [Derived] Krolewiecki A, Enbiale W, Gandasegui J, van Lieshout L, Kepha S, Messa Junior A, Bengtson M, Gelaye W, Escola V, Martinez-Valladares M, Cambra-Pelleja M, Algorta J, Marti-Soler H, Fleitas P, Ballester MR, Doyle SR, Williams NA, Legarda A, Mandomando I, Mwandawiro C, Munoz J. An adaptive phase II/III safety and efficacy randomized controlled trial of single day or three-day fixed-dose albendazole-ivermectin co-formulation versus albendazole for the treatment of Trichuris trichiura and other STH infections. ALIVE trial protocol. Gates Open Res. 2022 May 5;6:62. doi: 10.12688/gatesopenres.13615.1. eCollection 2022. PMID 36540062

RESULTS

PARTICIPANT FLOW:
Groups:
- Albendazole: Single dose of Albendazole 400mg
- Single Dose Albendazole-Ivermectin Fixed Dose Co-formulation (FDCx1): Single dose 400mg Albendazole- 9mg Ivermectin for participants <45 kg of body weight Single dose 400mg Albendazole- 18mg Ivermectin for participants >= 45 kg of body weight
- Daily Dose of Albendazole-Ivermectin FIxed Dose Co-formulation for Three Consecutive Days (FDCx3): Daily dose of 400mg Albendazole- 9mg Ivermectin for 3 consecutive days for participants <45 kg of body weight Daily dose of 400mg Albendazole- 18mg Ivermectin for 3 consecutive days for participants >= 45 kg of body weight
Period: Phase II
Arm/Group | Albendazole | Single Dose Albendazole-Ivermectin Fixed Dose Co-formulation (FDCx1) | Daily Dose of Albendazole-Ivermectin FIxed Dose Co-formulation for Three Consecutive Days (FDCx3)
Started | 30 | 51 | 54
Received Any Study Drug After Randomization | 27 | 50 | 51
Completed | 24 | 48 | 51
Not Completed | 6 | 3 | 3
Not completed — Eligibility criteria | 0 | 1 | 0
Not completed — Withdrawal by Subject | 6 | 2 | 3
Period: Phase III
Arm/Group | Albendazole | Single Dose Albendazole-Ivermectin Fixed Dose Co-formulation (FDCx1) | Daily Dose of Albendazole-Ivermectin FIxed Dose Co-formulation for Three Consecutive Days (FDCx3)
Started | 213 | 330 | 323
Received Any Study Drug After Randomization | 213 | 330 | 323
Completed | 206 | 326 | 319
Not Completed | 7 | 4 | 4
Not completed — Withdrawal by Subject | 6 | 4 | 4
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The variation in participant numbers is attributed to the differing allocation ratios for each infection. Specifically, the allocation rate was 1:2:2 for Trichuris, 1:1:1 for hookworm, and 2:5:5 for S. stercoralis, reflecting the study's design for each pathogen
Groups:
- Total: Total of all reporting groups
Arm/Group | Albendazole | Single Dose Albendazole-Ivermectin Fixed Dose Co-formulation (FDCx1) | Daily Dose of Albendazole-Ivermectin FIxed Dose Co-formulation for Three Consecutive Days (FDCx3) | Total
Number analyzed (Participants) | 243 | 381 | 377 | 1001
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Phase II (n=135) and Phase III (n=866) data are shown separately
  Years
    Phase II: number analyzed (Participants) | 30 | 51 | 54 | 135
    Phase II | 9.0 (2.55) | 8.9 (2.66) | 9.2 (2.74) | 9.1 (2.65)
    Phase III: number analyzed (Participants) | 213 | 330 | 323 | 866
    Phase III | 11.4 (3.08) | 11.2 (3.05) | 11.3 (3.24) | 11.3 (3.13)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Phase II (n=135) and Phase III (n=866) data are shown separately
  Participants
    Phase II: number analyzed (Participants) | 30 | 51 | 54 | 135
    Phase II: Female | 20 | 28 | 31 | 79
    Phase II: Male | 10 | 23 | 23 | 56
    Phase III: number analyzed (Participants) | 213 | 330 | 323 | 866
    Phase III: Female | 113 | 165 | 179 | 457
    Phase III: Male | 100 | 165 | 144 | 409
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Phase II (n=135) and Phase III (n=866) data are shown separately
  Participants
    Phase II: number analyzed (Participants) | 30 | 51 | 54 | 135
    Phase II: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Phase II: Asian | 0 | 0 | 0 | 0
    Phase II: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Phase II: Black or African American | 30 | 51 | 54 | 135
    Phase II: White | 0 | 0 | 0 | 0
    Phase II: More than one race | 0 | 0 | 0 | 0
    Phase II: Unknown or Not Reported | 0 | 0 | 0 | 0
    Phase III: number analyzed (Participants) | 213 | 330 | 323 | 866
    Phase III: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Phase III: Asian | 0 | 0 | 0 | 0
    Phase III: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Phase III: Black or African American | 213 | 330 | 323 | 866
    Phase III: White | 0 | 0 | 0 | 0
    Phase III: More than one race | 0 | 0 | 0 | 0
    Phase III: Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: Phase II (n=135) and Phase III (n=866) data are shown separately
  Participants
    Ethiopia: number analyzed (Participants) | 96 | 107 | 104 | 307
    Ethiopia: Phase II | 0 | 0 | 0 | 0
    Ethiopia: Phase III | 96 | 107 | 104 | 307
    Kenya: number analyzed (Participants) | 114 | 209 | 209 | 532
    Kenya: Phase II | 30 | 51 | 54 | 135
    Kenya: Phase III | 84 | 158 | 155 | 397
    Mozambique: number analyzed (Participants) | 33 | 65 | 64 | 162
    Mozambique: Phase II | 0 | 0 | 0 | 0
    Mozambique: Phase III | 33 | 65 | 64 | 162
Number of subjects positive for infection with T. trichiura [Count of Participants; unit: Participants] — Population: Phase II (n=135) and Phase III (n=866) data are shown separately.
  Participants
    Phase II: number analyzed (Participants) | 30 | 51 | 54 | 135
    Phase II | 30 | 51 | 54 | 135
    Phase III: number analyzed (Participants) | 213 | 330 | 323 | 866
    Phase III | 101 | 200 | 200 | 501
Eggs per gram (EPG) detected by Kato-Katz technique in participants infected with T. trchiura [Geometric Mean (Standard Deviation); unit: Eggs per gram of stool] — Population: The population corresponds to those infected at baseline with T. trichiura (n=636).
  Measure Analysis Population Description: Phase II (n=135) and Phase III (n=501) data are shown separately
  Eggs per gram of stool
    Phase II: number analyzed (Participants) | 30 | 51 | 54 | 135
    Phase II | 113.0 (1.2) | 137.4 (1.5) | 159.4 (1.4) | 139.6 (1.4)
    Phase III: number analyzed (Participants) | 101 | 200 | 200 | 501
    Phase III | 128.0 (1.5) | 124.2 (1.4) | 121.6 (1.5) | 123.9 (1.5)
Number of subjects positive for infection with Hookworms [Count of Participants; unit: Participants] — Population: Phase II (n=135) and Phase III (n=866) data are shown separately.
  Participants
    Phase II: number analyzed (Participants) | 30 | 51 | 54 | 135
    Phase II | 2 | 4 | 4 | 10
    Phase III: number analyzed (Participants) | 213 | 330 | 323 | 866
    Phase III | 106 | 124 | 120 | 350
Eggs per gram (EPG) detected by Kato-Katz technique in participants infected with hookworm [Geometric Mean (Standard Deviation); unit: Eggs per gram of stool] — Population: Measure Analysis Population Description: The population corresponds to those infected at baseline with hookworms (n=360).
  Measure Analysis Population Description: Phase II (n=10) and Phase III (n=350) data are shown separately
  Eggs per gram of stool
    Phase II: number analyzed (Participants) | 2 | 4 | 4 | 10
    Phase II | 42.6 (0.2) | 527.3 (1.5) | 93.0 (2.3) | 159.2 (1.9)
    Phase III: number analyzed (Participants) | 106 | 124 | 120 | 350
    Phase III | 116.6 (1.3) | 118.2 (1.3) | 112.9 (1.4) | 115.9 (1.3)
Number of subjects positive for infection with S. stercoralis [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Phase II (n=135) and Phase III (n=866) data are shown separately
  Participants
    Phase II: number analyzed (Participants) | 30 | 51 | 54 | 135
    Phase II | 0 | 4 | 3 | 7
    Phase III: number analyzed (Participants) | 213 | 330 | 323 | 866
    Phase III | 16 | 40 | 41 | 97

OUTCOME MEASURES:

1. Primary Outcome: Cure Rate for T. Trichiura (CR)
Description: For Trichuris trichiura, the cure rate is defined as the proportion of participants who test negative for T. trichiura eggs in the Kato-Katz fecal examination on day 21 post-treatment, relative to the total number of participants infected at baseline (n=636).
Time Frame: 21 days
Population: Intention to treat population infected with Trichuris trichiura from both Phase II and Phase III of the study (n=636).
  A separate efficacy analysis by phase was not conducted, as the protocol specifies that the required sample size for this outcome is derived from all participants infected with T. trichiura at baseline, combining those from Phase II and Phase III.
Measure: Count of Participants; unit: Participants
Arm/Group | Albendazole | Single Dose Albendazole-Ivermectin Fixed Dose Co-formulation (FDCx1) | Daily Dose of Albendazole-Ivermectin FIxed Dose Co-formulation for Three Consecutive Days (FDCx3)
Number analyzed (Participants) | 131 | 251 | 254
Participants | 47 | 208 | 247
Statistical Analysis 1: Comparison: Albendazole vs Single Dose Albendazole-Ivermectin Fixed Dose Co-formulation (FDCx1); pairwise comparisons of cure rates within the three study groups, considering an overall significance level of 0.05. To account for multiple testing, a Bonferroni correction was applied, resulting in an adjusted significance level of 0.0167; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Albendazole vs Daily Dose of Albendazole-Ivermectin FIxed Dose Co-formulation for Three Consecutive Days (FDCx3); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Single Dose Albendazole-Ivermectin Fixed Dose Co-formulation (FDCx1) vs Daily Dose of Albendazole-Ivermectin FIxed Dose Co-formulation for Three Consecutive Days (FDCx3); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel

2. Primary Outcome: Frequency of Related Adverse Events
Description: Proportions of participants presenting at least one treatment-related adverse event by arm
Time Frame: 21 days postreatment
Population: Intention-to-Treat (ITT) population from both Phase II and Phase III (n = 1001), regardless of baseline infection type (T. trichiura, hookworms, or S. stercoralis).
Measure: Count of Participants; unit: Participants
Arm/Group | Albendazole | Single Dose Albendazole-Ivermectin Fixed Dose Co-formulation (FDCx1) | Daily Dose of Albendazole-Ivermectin FIxed Dose Co-formulation for Three Consecutive Days (FDCx3)
Number analyzed (Participants) | 243 | 381 | 377
Participants
  ITT Phase II and Phase III | 34 | 75 | 88
  ITT Phase II: number analyzed (Participants) | 30 | 51 | 54
  ITT Phase II | 3 | 8 | 10
  ITT Phase III: number analyzed (Participants) | 213 | 330 | 323
  ITT Phase III | 31 | 67 | 78

3. Secondary Outcome: Egg Reduction Rate for T. Trichiura (ERR)
Description: The Egg Reduction Rate (ERR) is defined as the percentage reduction in the geometric mean (GM) of eggs per gram (EPG) of feces from baseline to post-treatment.
Time Frame: 21 days
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Percentage of reduction
Arm/Group | Albendazole | Single Dose Albendazole-Ivermectin Fixed Dose Co-formulation (FDCx1) | Daily Dose of Albendazole-Ivermectin FIxed Dose Co-formulation for Three Consecutive Days (FDCx3)
Number analyzed (Participants) | 131 | 251 | 254
Percentage of reduction | 83.4 [73.7 to 89.8] | 99.2 [98.9 to 99.5] | 99.9 [99.8 to 99.9]

4. Secondary Outcome: Cure Rate for for Hookworm (CR)
Description: For hookworm, the cure rate is defined as the proportion of participants who test negative for hookworm eggs in the Kato-Katz fecal examination on day 21 post-treatment, relative to the total number of participants infected at baseline in Phase III (n=350).
Time Frame: 21 days
Population: Intention to treat population infected with hookworm from Phase III of the study (n=350).
  A separate efficacy analysis by phase was not conducted, as the protocol specifies that the required sample size for this outcome is derived exclusively from participants infected with hookworms at baseline in Phase III.
Measure: Count of Participants; unit: Participants
Arm/Group | Albendazole | Single Dose Albendazole-Ivermectin Fixed Dose Co-formulation (FDCx1) | Daily Dose of Albendazole-Ivermectin FIxed Dose Co-formulation for Three Consecutive Days (FDCx3)
Number analyzed (Participants) | 106 | 124 | 120
Participants | 69 | 99 | 114
Statistical Analysis 1: Comparison: Albendazole vs Daily Dose of Albendazole-Ivermectin FIxed Dose Co-formulation for Three Consecutive Days (FDCx3); Pairwise comparisons of cure rates were conducted between Albendazole and FDCx3, as well as FDCx1 and FDCx3, but not between Albendazole and FDCx1, since both contain the same dose regimen of the active drug. An overall significance level of 0.05 was considered, and to account for multiple testing, a Bonferroni correction was applied; Test type: Superiority; p < 0.0001, Mantel Haenszel
Statistical Analysis 2: Comparison: Single Dose Albendazole-Ivermectin Fixed Dose Co-formulation (FDCx1) vs Daily Dose of Albendazole-Ivermectin FIxed Dose Co-formulation for Three Consecutive Days (FDCx3); [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0007, Cochran-Mantel-Haenszel

5. Secondary Outcome: Egg Reduction Rate for Hookworm (ERR)
Description: as for outcome 3
Time Frame: 21 days
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Percentage of reduction
Arm/Group | Albendazole | Single Dose Albendazole-Ivermectin Fixed Dose Co-formulation (FDCx1) | Daily Dose of Albendazole-Ivermectin FIxed Dose Co-formulation for Three Consecutive Days (FDCx3)
Number analyzed (Participants) | 106 | 124 | 120
Percentage of reduction | 97.8 [96.6 to 98.7] | 99.0 [98.2 to 99.4] | 99.8 [99.5 to 99.9]

6. Secondary Outcome: Cure Rates for for S. Stercoralis
Description: For S. stercoralis, the cure rate is defined as the proportion of participants who test negative for S. stercoralis larvae in the Baermann tesi on day 21 post-treatment, relative to the total number of participants infected at baseline in Phase III (n=97).
Time Frame: 21 days
Population: Intention to treat population infected with S. stercoralis from Phase III of the study (n=97).
  A separate efficacy analysis by phase was not conducted, as the protocol specifies that the required sample size for this outcome is derived exclusively from participants infected with S. stercoralis at baseline in Phase III.
Measure: Count of Participants; unit: Participants
Arm/Group | Albendazole | Single Dose Albendazole-Ivermectin Fixed Dose Co-formulation (FDCx1) | Daily Dose of Albendazole-Ivermectin FIxed Dose Co-formulation for Three Consecutive Days (FDCx3)
Number analyzed (Participants) | 16 | 40 | 41
Participants | 13 | 38 | 41

7. Secondary Outcome: Cure Rate for T. Trichiura (CR) by qPCR
Description: For Trichuris trichiura, the cure rate is defined as the proportion of participants who test negative by qPCR (Ct-value>35) on day 21 post-treatment, relative to the total number of participants that were positves at baseline by Kato-Katz and qPCR (n=534).
Time Frame: 21 days
Population: For Trichuris trichiura, the cure rate is defined as the proportion of participants who test negative by qPCR (Ct-value>35) on day 21 post-treatment, relative to the total number of participants that were positves at baseline by Kato-Katz and qPCR (n=534).
Measure: Count of Participants; unit: Participants
Arm/Group | Albendazole | Single Dose Albendazole-Ivermectin Fixed Dose Co-formulation (FDCx1) | Daily Dose of Albendazole-Ivermectin FIxed Dose Co-formulation for Three Consecutive Days (FDCx3)
Number analyzed (Participants) | 110 | 203 | 221
Participants | 55 | 152 | 188
Statistical Analysis 1: Comparison: Albendazole vs Single Dose Albendazole-Ivermectin Fixed Dose Co-formulation (FDCx1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Albendazole vs Daily Dose of Albendazole-Ivermectin FIxed Dose Co-formulation for Three Consecutive Days (FDCx3); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Single Dose Albendazole-Ivermectin Fixed Dose Co-formulation (FDCx1) vs Daily Dose of Albendazole-Ivermectin FIxed Dose Co-formulation for Three Consecutive Days (FDCx3); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel

8. Secondary Outcome: To Evaluate the Frequency of Known ALB Resistant Alleles in Hookworm and T. Trichiura in the Three Treatment Arms Before and After Treatment.
Description: The original objective as per the protocol was to "To evaluate the frequency of known ALB resistant alleles in hookworm and T. trichiura in the three treatment arms before and after treatment" with the endpoint being "Evaluation of genotypic albendazole resistance in the three arms." This objective was based on the hypothesis that mutations at codons 167, 198, and 200 of the beta-tubulin gene of Trichuris trichiura were associated with resistance. However, since this time, it has become increasingly evident, based on research from us (PMID: 35895348, 39546832, 34563247) and others, that this hypothesis is no longer supported, and that the genetic determinants of resistance in T. trichiura are yet to be discovered. Therefore, we have begun evaluating, using whole genome sequencing, other genetic variants and their association with poor treatment response. This research is exploratory and ongoing. Therefore, the original outcome as defined in the protocol could not be assessed.
Time Frame: 21 days
Population: Although samples were collected from participants, they were not analyzed and will not be analyzed in the future, as emerging scientific evidence has invalidated the hypothesis.
Arm/Group | Albendazole | Single Dose Albendazole-Ivermectin Fixed Dose Co-formulation (FDCx1) | Daily Dose of Albendazole-Ivermectin FIxed Dose Co-formulation for Three Consecutive Days (FDCx3)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: For the safety evaluation on treatment days, participants stayed at the sites for 3 h after drug administration.Safety was also actively monitored on days 1, 2, 7, and 21 after taking the medication.
Description: Adverse events were reported for the intention-to-treat (ITT) population comprising participants from both Phase II and Phase III (n = 1001), regardless of baseline infection type (T. trichiura, hookworms, or S. stercoralis). All events were documented systematically following treatment administration.
Arm/Group | Albendazole | Single Dose Albendazole-Ivermectin Fixed Dose Co-formulation (FDCx1) | Daily Dose of Albendazole-Ivermectin FIxed Dose Co-formulation for Three Consecutive Days (FDCx3)
All-Cause Mortality (participants affected / at risk) | 0/243 | 0/381 | 0/377
Serious Adverse Events (participants affected / at risk) | 0/243 | 0/381 | 0/377
Other Adverse Events (participants affected / at risk) | 50/243 | 99/381 | 107/377
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albendazole (N=243) | Single Dose Albendazole-Ivermectin Fixed Dose Co-formulation (FDCx1) (N=381) | Daily Dose of Albendazole-Ivermectin FIxed Dose Co-formulation for Three Consecutive Days (FDCx3) (N=377)
Abdominal pain (Gastrointestinal disorders) | 23 (24) | 52 (60) | 47 (52)
Headache (Nervous system disorders) | 7 (7) | 20 (21) | 14 (18)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 17 (17) | 12 (14)
Vomiting (Gastrointestinal disorders) | 4 (4) | 10 (10) | 12 (15)
Nausea (Gastrointestinal disorders) | 2 (2) | 6 (6) | 17 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 10 (10)
Parasitic gastroenteritis (Gastrointestinal disorders) | 3 (5) | 3 (3) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 5 (5)
Upper respiratory track infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 2 (2)

LIMITATIONS AND CAVEATS:
Pre-specified sample size for evaluating the efficacy of FDCx1 and FDCx3 versus albendazole for the treatment of S. stercoralis was not met, the available data were collected and summarized descriptively. These results are reported in Outcome Measure 6. However, due to the insufficient sample size, no formal statistical analysis was performed, and the findings are presented for descriptive purposes only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-01-21): https://cdn.clinicaltrials.gov/large-docs/91/NCT05124691/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT05124691/SAP_001.pdf